CLINICAL TRIAL: NCT04733911
Title: Recovery Kinetics Following Three Exercise-induced Muscle Damage Protocols in Adult Males
Brief Title: Recovery Kinetics Following Eccentric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Recovery-Eccentrics-UTH
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Muscle Damage
Keywords: muscle damage; oxidative stress; Eccentric exercise; Neuromuscular fatigue; Recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Eccentric 75 (Experimental): Participants in this arm will perform an eccentric exercise protocol consisted of 75 eccentric repetetions on an isokinetic dynamometer.
  Interventions: Other: 75 eccentric contractions
- Eccentric 150 (Experimental): Participants in this arm will perform an eccentric exercise protocol consisted of 150 eccentric repetetions on an isokinetic dynamometer.
  Interventions: Other: 150 eccentric contractions
- Eccentric 300 (Experimental): Participants in this arm will perform an eccentric exercise protocol consisted of 300 eccentric repetetions on an isokinetic dynamometer.
  Interventions: Other: 300 eccentric contractions
- Control (No Intervention): Participants in this arm will receive no intervention.

INTERVENTIONS:
Other: 75 eccentric contractions — An acute bout of eccentric exercise will be performed on an isokinetic dynamometer, including 5 sets of 15 repetitions, with 30 sec rest intervals,at 60 degrees/sec.
  Arms: Eccentric 75
Other: 150 eccentric contractions — An acute bout of eccentric exercise will be performed on an isokinetic dynamometer, including 10 sets of 15 repetitions, with 30 sec rest intervals,at 60 degrees/sec.
  Arms: Eccentric 150
Other: 300 eccentric contractions — An acute bout of eccentric exercise will be performed on an isokinetic dynamometer, including 20 sets of 15 repetitions, with 30 sec rest intervals,at 60 degrees/sec.
  Arms: Eccentric 300

SUMMARY:
The aim of this study will be to investigate the recovery kinetics of neuromuscular fatigue, muscle microtrauma indicators, performance and oxidative stress factors after three different exercise induced muscle damage (EIMD) protocols in adult Males. Also, this study will determine the comparison among three different eccentric protocols in neuromuscular fatigue, muscle microtrauma indicators, performance and oxidative stress factors. The eccentric protocols will be differentiated in training volume and specifically in the eccentric repetitions in isokinetic dynamometer.

DETAILED DESCRIPTION:
It is known that eccentric exercise induces muscle microtrauma. Also, eccentric type of exercise are associated with inflammatory response. The leukocytes and the immune cells during the phagocytosis process alter the redox status causing secondary muscle damage to the muscle tissue and also increase oxidative stress concentration. Despite of the existence of studies that examine the muscle damage indicators, inflammatory response, performance and neuromuscular fatigue and oxidative stress concentrations after eccentric exercise, however no studies are detected in order to compare the differences among three eccentric protocols. The eccentric protocols will be differentiated in training volume and specifically in the eccentric repetitions in isokinetic dynamometer. Specifically, a randomized, fourth-trial, cross-over, repeated measures design will be applied. Healthy male adults (age 18-30 years) will participate in the present study. Also, it is considered necessary that the participants will not suffer from any musculoskeletal injuries that will limit their ability to perform the exercise protocols. Also the participants will not be smokers and will not consume alcohol and nutritional supplements.

In the first phase all participants will sign an informed consent form after they will be informed about all benefits and risks of this study and they will sign a recent historical of musculoskeletal injury or illness form. Subsequently, fasting blood samples will be collected by venipuncture using a disposable needle (20-gauge) in order to measure muscle damage markers (CK), inflammation markers (WBC) and oxidative stress markers (TBARS, PC, GSH, ΤΑC, CAT, UA). After, delayed onset muscle soreness (DOMS) in the knee flexors (KF) and extensors (KE) of both limbs, body weight (BW), height and body composition (DXA method) will be measured in the lab. Completing the first phase, participants will be instructed by a dietitian how to record a 5 days diet recalls estimating the energy intake during the trials will be the same. The knee range of motion (KJRM) will be determined by the use of a goniometer, 24 hours after (second phase). The counter movement jump (CMJ) will be evaluated on a force platform using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg. During the CMJ will be measured the jump height (cm), the ground reaction force (N), the peak and mean power (W/kg), the vertical stiffness (Kvert, N/m/kg) and the peak rate of force development (RFD, N/s), while at the same time will be evaluated the change in peak and mean normalized EMG during the eccentric and concentric phases of the counter movement jump, for the vastus medialis (VM) and vastus lateralis muscles. Electromyography data will be collected wirelessly at 2.000 Hz using a Myon MA-320 EMG system. The peak eccentric and concentric isokinetic torque of the knee flexors and extensors, in both limbs will be evaluated on an isokinetic dynamometer at 60°/sec. Also, the isometric peak torque of the knee extensors will be evaluated at 65° in both limbs. Finally, Open-circuit spirometry will be utilized for assessment of maximal oxygen consumption (VO2max) using an automated online pulmonary gas exchange system via breath-by-breath analysis during a graded exercise testing on a treadmill.

96 hours after, the participants are going to perform one of the three eccentric protocols randomly, on an isokinetic dynamometer. The eccentric protocol will be performed on a different limb for each trial. The ECC 75 trial will include 75 eccentric maximum repetitions (5 sets, 15 reps/set and recovery period: 30sec.) at 60°/sec. The ECC 150 trial will include 150 eccentric maximum repetitions (10 sets, 15 reps/set and recovery period: 30sec.) at 60°/sec. The ECC 300 trial will include 300 eccentric maximum repetitions (20 sets, 15 reps/set and recovery period: 30sec.) at 60°/sec. The DOMS indicator in the knee flexors (KF) and extensors (KE) of both limbs and the KJRM will be evaluated immediately after each protocol. Also, the (CMJ) will be evaluated on a force platform using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg. During the CMJ will be measured the jump height (cm), the ground reaction force (N), the peak and mean power (W/kg), the vertical stiffness (Kvert, N/m/kg) and the peak rate of force development (RFD, N/s), while at the same time will be evaluated the change in peak and mean normalized EMG during the eccentric and concentric phases of the counter movement jump, for the vastus medialis (VM) and vastus lateralis muscles. Electromyography data will be collected wirelessly at 2.000 Hz using a Myon MA-320 EMG system. In addition, the peak eccentric and concentric isokinetic torque of the knee flexors and extensors, in both limbs will be evaluated on an isokinetic dynamometer at 60o/sec. Also, the isometric peak torque of the knee extensors will be evaluated at 65o in both limbs. All the above markers will be evaluated 24, 48 and 192 hours post eccentric protocol, however at these time points, fasting blood samples (20ml) will be collected in order to estimate hematological and biochemical indicators. Α 2 - week washout period will be adapted among trials. After, the participants will perform the process until they complete the trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years
* Body Mass Index between 18.5-24.9 kg/m*m
* Free of chronic diseases
* Free of musculoskeletal injury
* participants should be non-smokers

Exclusion Criteria:

* Musculoskeletal injury
* Chronic disease
* Use of alcohol, caffeine and any type of nutritional supplements or medication before (≥ 6 months) and throughout the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in white blood cell count | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  White blood cell count will be measured using an automatic blood analyzer
Change in catalase activity | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Concentration of catalase will be measured in red blood cells
Change in uric acid in plasma | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  concentration of uric acid will be measured in plasma
Change in protein carbonyls in blood | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Concentration of protein carbonyls will be measured in red blood cells
Change in total antioxidant capacity | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  total antioxidant capacity will be measured in serum
Change in reduced glutathione in blood | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Concentration of oxidized glutathione will be measured in red blood cells
Change in thiobarbituric acid reactive substances | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Thiobarbituric acid will be measured in plasma
Change in Creatine kinase in blood | At baseline, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Creatine kinase will be measured in plasma
Change in countermovement jump height | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  Countermovement jump height will be measured using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the jump height data for each leg.
Change in ground reaction force (GRF) during countermovement jump test | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  The ground reaction force will be measured using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the GRF data for each leg.
Change in peak power during countermovement jump test | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  The peak power will be measured using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the peak power data for each leg.
Change in mean power during countermovement jump test | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  The mean power will be measured using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the mean power data for each leg.
Change in vertical stifness during countermovement jump test | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  The vertical stiffness will be measured using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of vertical stifness data for each leg.
Change in peak rate of force develpemnt during countermovement jump test | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  The Peak rate of force development will be measured using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the Peak RFD data for each leg.
Change in peak normalized EMG during the eccentric and concentric phases of the counter movement jump | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  Electromyography data will be collected wirelessly at 2.000 Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus medialis (VM) and vastus lateralis muscles.
Change in mean normalized EMG during the eccentric and concentric phases of the counter movement jump | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  Electromyography data will be collected wirelessly at 2.000 Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus medialis (VM) and vastus lateralis muscles.
Change in knee range of motion | At baseline, at 1 hour and 24, 48 and 192 hours following the eccentric exercise protocol.
  Knee range of motion will be measured by goniometer
Change in eccentric isokinetic knee extensors peak torque | At baseline, 1 hour, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Eccentric isokinetic knee extensors peak torque will be assessed on an isokinetic dynamometer
Change in concentric isokinetic knee extensors peak torque | At baseline, 1 hour, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Concentric isokinetic knee extensors peak torque will be assessed on an isokinetic dynamometer
Change in eccentric isokinetic knee flexors peak torque | At baseline, 1 hour, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Eccentric isokinetic knee flexors peak torque will be assessed on an isokinetic dynamometer
Change in concentric isokinetic knee flexors peak torque | At baseline, 1 hour, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Concentric Iisokinetic knee flexors peak torque will be assessed on an isokinetic dynamometer
Change in isometric peak torque | At baseline, 1 hour, at 24, 48 and 192 hours following the eccentric exercise protocol.
  The isometric peak torque will be assessed on an isokinetic dyanmometer
Change in fatigue index of isometric torque during 10 second | At baseline, 1hour, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Fatigue rate during MVIC will be estimated through the percent drop of peak torque between the first and the last three seconds of a 10-secong maximal isometric contraction.
Change in delayed onset of muscle soreness (DOMS) in the knee flexors (KF) and extensors (KE) of both limbs | At baseline, 1 hour, at 24, 48 and 192 hours following the eccentric exercise protocol.
  Muscle soreness (KF and KE) will be assessed during palpation of the muscle belly and the distal region

SECONDARY OUTCOMES:
Body weight | At baseline
  Body weight will be measured on a beam balance with stadiometer
Body height | At baseline
  Body height will be measured on a beam balance with stadiometer
Body fat | At baseline
  Body fat will be measured by using Dual-emission X-ray absorptiometry
Dietary intake | Over a 5 -day period at baseline
  Dietary intake will be assessed using 5 -day diet recalls
Maximal oxygen consumption (VO2max) | At baseline
  Maximal oxygen consumption will be measured by open circuit spirometry via breath by breath method

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, Prof, Study Director — University of Thessaly
Locations (1):
- University o Thessaly, School of Physical Education and Sports Science, Trikala, Greece